CLINICAL TRIAL: NCT01151501
Title: Noninvasive Positive Pressure Ventilation for Early Extubation of Acute Hypoxemic Respiratory Failure
Acronym: NPPV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We anticipated that we could not complete this study.
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Zujin Luo, MD, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BeijingCYH-ICU-000
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: acute hypoxemic respiratory failure; intermittent positive-pressure ventilation; noninvasive positive pressure ventilation; ventilator weaning
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- noninvasive positive pressure ventilation (Experimental)
  Interventions: Device: noninvasive positive pressure ventilation

INTERVENTIONS:
Device: noninvasive positive pressure ventilation — Patients in whom the spontaneous breathing trial fail and in whom exclusion criteria are not present during this period were randomly allocated. Patients who are randomized to NPPV goup will be extubated and non-invasive ventilation (BiPAP Vision, Respironics Inc., Murrysville，Pennsylvania) will be delivered immediately after extubation using spontaneous/timed (S/T) mode. Expiratory positive airways pressure (PEEP) was initially set at 4 cmH2O and gradually increased to 6-8 cmH2O or more；and fraction of inspired oxygen (FiO2) was set to achieve pulse oximeter oxygen saturation (SpO2) >92% in cooperation with PEEP. On condition that tidal volume is no less than 6ml/kg，continuous positive airway pressure (CPAP) is permitted to apply，in which the adjusting procedures of CPAP and FiO2 is similar with PEEP and FiO2 in S/T mode. NPPV is terminated When patients can spontaneously breath oxygen provided by a Venturi device at FiO2≤0.35 for more than 24 hours with SpO2>92%.

SUMMARY:
Acute hypoxaemic respiratory failure (AHRF) refers to pathological states in which arterial blood oxygenation is severely impaired，and which need invasive positive pressure ventilation (IPPV) as respiratory support technique in most cases.However，IPPV carries well-known risks of complications such as ventilator induced lung injury (VILI) or ventilator associated pneumonia (VAP)，and the incidence of which is increased as the prolongation of IPPV so as to lead to higher mortality rate. Consequently，early extubation is extraordinarily necessary.

More recently, NPPV has shown to shorten the duration of IPPV，reduce the mortality and morbidity rates in patients with chronic obstructive pulmonary disease (COPD). Despite this evidence, the efficacy of NPPV in patients with AHRF has not been evidenced. However，NPPV has been shown to provide adequate ventilation and oxygenation，and reduce inspiratory muscle effort，neuromuscular drive，and dyspnea scores. Moreover，to some patints，NPPV is similar with IPPV in providing oxygenation.

The duration of weaning is from the first day a patient met standard criteria for weaning readiness to the time of successful extubation (lasting at least 48 h)，which represents 40-50% of the total duration of IPPV.As a result，duration of IPPV would be shortened if that of weaning was shortened.

The investigators hypothesized that in mechanical ventilated patients with AHRF who met standard criteria for weaning readiness and suffer failure of spontaneous breathing trial, use of NPPV for early extubation, providing adequate ventilation and oxygenation, would shorten the duration of IPPV as the primary end-point variable, thereby reduce the incidence of complication and mortality rates. Accordingly, the investigators conducted a prospective，randomized clinical trial to assess the efficacy of this strategy compared with the conventional-weaning approach.

ELIGIBILITY:
Inclusion Criteria:

* Orotracheal intubation
* Arterial oxygen tension (PaO2)<60mmHg（venturi mask，FiO2=0.5），and arterial carbon dioxide tension(PaCO2)≤45mmHg；
* Meeting standard criteria for weaning readiness
* Suffering failure of spontaneous breathing trial.

Exclusion Criteria:

* Age<18
* Duration of invasive positive pressure ventilation<48h
* Tracheotomy
* Percentage of cuff leak volume in tidal volume<15.5%
* Unable to spontaneously clear secretions from their airway
* Recent oral，nasal，facial or cranial trauma or surgery
* Recent gastric or esophageal surgery
* Active upper gastro-intestinal bleeding
* Severe abdominal distension
* Lack of co-operation
* Chronic respiratory disease such as chronic obstructive pulmonary disease，asthma，interstitial lung disease,etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Duration of invasive positive pressure ventilation | two year

SECONDARY OUTCOMES:
Incidence of ventilator associated pneumonia | two year
Intensive care unit mortality | two years
Hospital mortality | two years
90-day survival after entry | two years

CONTACTS AND LOCATIONS:
Overall Officials: Wang Chen, MD, Study Chair — Beijing Chao Yang Hospital; Zhan Q Yuan, MD, Study Director — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chao Yang Hospital, Beijing, Beijing Municipality, China